CLINICAL TRIAL: NCT00445770
Title: A Randomized, Double-Blind, Multicenter, Comparative Study Evaluating the Efficacy and Safety of Etanercept and Methotrexate in Japanese Subjects With Active Rheumatoid Arthritis
Brief Title: Study Evaluating the Efficacy and Safety of Etanercept and Methotrexate in Japanese Subjects With Rheumatoid Arthritis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0881A1-315; B1801002
Record Dates: First submitted 2007-03-08; First posted 2007-03-09 (Estimated); Results first posted 2011-08-05 (Estimated); Last update posted 2011-08-15 (Estimated); Status verified 2011-08

CONDITIONS: Arthritis, Rheumatoid
Keywords: Rheumatoid Arthritis; Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid; Arthritis | interventions — Etanercept; Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 (Experimental)
  Interventions: Drug: Etanercept
- 2 (Experimental)
  Interventions: Drug: Etanercept
- 3 (Active Comparator)
  Interventions: Drug: Methotrexate

INTERVENTIONS:
Drug: Etanercept — 10 mg twice weekly, subcutaneous injection for 52 weeks
  Arms: 1
Drug: Etanercept — 25 mg, twice weekly, subcutaneous injection for 52 weeks
  Arms: 2
Drug: Methotrexate — up to 8 mg per week, oral dosing for 52 weeks
  Arms: 3

SUMMARY:
The purpose of this study is to examine the effects of etanercept (10 mg and 25 mg) compared with methotrexate (up to 8 mg per week) on the slowing of joint destruction.

ELIGIBILITY:
Inclusion Criteria:

* Must be Japanese and live in Japan
* Must be age 20 to 75 years
* Diagnosed less than or equal to 10 years from time of first visit

Exclusion Criteria:

* Anyone who has received etanercept or TNF-inhibitors such as infliximab or adalimumab in the past
* Patient with other rheumatic diseases or conditions that could predispose the patient to infection
* Pregnant or lactating women

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 550 (Actual)
Dates: Start 2006-07; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (35):
- Japan (35):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Goshogawara, Aomori
  - Pfizer Investigational Site, Asahi, Chiba
  - Pfizer Investigational Site, Matsuyama, Ehime
  - Pfizer Investigational Site, Fukui-shi, Fukui
  - Pfizer Investigational Site, Fukuoka, Fukuoka
  - Pfizer Investigational Site, Iizuka, Fukuoka
  - Pfizer Investigational Site, Kurume, Fukuoka
  - Pfizer Investigational Site, Munakata, Fukuoka
  - Pfizer Investigational Site, Takasaki, Gunma
  - Pfizer Investigational Site, Hiroshima, Hiroshima
  - Pfizer Investigational Site, Asahikawa, Hokkaido
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Kakogawa, Hyōgo
  - Pfizer Investigational Site, Katoh, Hyōgo
  - Pfizer Investigational Site, Yūki, Ibaraki
  - Pfizer Investigational Site, Komatsu, Ishikawa-ken
  - Pfizer Investigational Site, Kagoshima, Kagoshima-ken
  - Pfizer Investigational Site, Kawasaki, Kanagawa
  - Pfizer Investigational Site, Sagamihara, Kanagawa
  - Pfizer Investigational Site, Yokohama, Kanagawa
  - Pfizer Investigational Site, Kumamoto, Kumamoto
  - Pfizer Investigational Site, Miyagi, Miyagi
  - Pfizer Investigational Site, Sendai, Miyagi
  - Pfizer Investigational Site, Hyūga, Miyazaki
  - Pfizer Investigational Site, Miyazaki, Miyazaki
  - Pfizer Investigational Site, Sasebo, Nagasaki
  - Pfizer Investigational Site, Ikoma, Nara
  - Pfizer Investigational Site, Kawagoe, Saitama
  - Pfizer Investigational Site, Tokorozawa, Saitama
  - Pfizer Investigational Site, Bunkyo-ku, Tokyo
  - Pfizer Investigational Site, Ōta-ku, Tokyo
  - Pfizer Investigational Site, Sumida-ku, Tokyo
  - Pfizer Investigational Site, Toyama, Toyama
  - Pfizer Investigational Site, Kato City Fujita Letter Higashiyama

REFERENCES:
- [Derived] Takeuchi T, Miyasaka N, Pedersen RD, Sugiyama N, Hirose T. Radiographic and clinical effects of 10 mg and 25 mg twice-weekly etanercept over 52 weeks in Japanese patients with active rheumatoid arthritis. Mod Rheumatol. 2021 Mar;31(2):319-325. doi: 10.1080/14397595.2020.1805142. Epub 2020 Sep 7. PMID 32735145
- [Derived] Takeuchi T, Miyasaka N, Pedersen R, Sugiyama N, Hirose T. Radiographic and clinical outcomes following etanercept monotherapy in Japanese methotrexate-naive patients with active rheumatoid arthritis. Mod Rheumatol. 2020 Mar;30(2):259-268. doi: 10.1080/14397595.2019.1589918. Epub 2019 Mar 29. PMID 30836801
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0881A1-315&StudyName=Study%20Evaluating%20the%20Efficacy%20and%20Safety%20of%20Etanercept%20and%20Methotrexate%20in%20Japanese%20Subjects%20with%20Rheumatoid%20Arthritis

RESULTS

PARTICIPANT FLOW:
Groups:
- Methotrexate: Participants received 4 milligrams (mg) up to 8 mg orally (2.0 mg capsules), once weekly for 52 weeks and subcutaneous (SC) placebo injections twice weekly
- Etanercept 10 mg: Participants received 10 mg SC twice weekly and oral placebo capsules once weekly for 52 weeks
- Etanercept 25 mg: Participants received 25 mg twice weekly SC and oral placebo capsules once weekly for 52 weeks
Period: Overall Study
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Started | 176 | 192 | 182
Completed | 123 | 157 | 151
Not Completed | 53 | 35 | 31
Not completed — Adverse Event | 9 | 15 | 19
Not completed — Lack of Efficacy | 38 | 13 | 6
Not completed — Lost to Follow-up | 0 | 2 | 0
Not completed — Other | 6 | 5 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg | Total
Number analyzed (Participants) | 176 | 192 | 182 | 550
Age Continuous [Mean (Standard Deviation); unit: years] | 50.40 (11.91) | 51.46 (12.21) | 51.81 (11.07) | 51.24 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 140 | 154 | 145 | 439
  Male | 36 | 38 | 37 | 111
modified Total Sharp Score (mTSS) [Mean (Standard Deviation); unit: scores on a scale] — mTSS=sum of erosion and JSN scores for 44 joints (16 per hand and 6 per foot). Total mTSS scores possible ranged from 0 (normal) to 448 (worst possible total score).
  scores on a scale | 43.01 (46.78) | 45.17 (38.75) | 41.98 (41.51) | 43.42 (42.28)
Erosion Score [Mean (Standard Deviation); unit: scores on a scale] — Joint erosion score: erosion severity in 44 joints (16 per hand and 6 per foot). Each joint scored according to surface area involved, from 0 (no erosion) to 5 (extensive bone loss from more than one half of articulating bone). Because each side of foot joint was graded, maximum erosion score for foot joint was 10. Thus, total erosion score possible ranged from 0 (no erosion) to 280 (worst possible total score).
  scores on a scale | 25.09 (26.30) | 26.66 (22.1) | 25.23 (23.88) | 25.69 (24.05)
Joint Space Narrowing (JSN) Score [Mean (Standard Deviation); unit: scores on a scale] — JSN score: severity of JSN in 42 joints (15 per hand and 6 per foot), including subluxation, scored from 0 (no/normal JSN) to 4 (complete loss of joint space, bony ankylosis, or luxation). Total JSN scores possible ranged from 0 (no/normal JSN) to 168 (worst possible total score).
  scores on a scale | 17.92 (21.93) | 18.50 (19.14) | 16.75 (19.11) | 17.73 (20.03)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) at Week 52
Description: mTSS = sum of erosion and JSN scores for 44 joints (16 per hand and 6 per foot). mTSS scores ranged from 0 (normal) to 448 (worst possible total score). Change = scores at observation minus score at Baseline. An increase in mTSS from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represents improvement.
Time Frame: Week 52
Population: Radiographic intent-to-treat (rITT) population: all participants who received at least 1 dose of the assigned test article and provided radiographic data for baseline and at least 1 post-baseline visit
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 171 | 190 | 181
Scores on a scale | 9.82 (1.16) | 5.19 (0.93) | 3.33 (0.73)
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; It was estimated that with 180 participants per group, there would be 81% power for the overall test. With this sample size and 0.05 (2-sided) type I error, there was 88% power to detect a 1.33 difference for the change of mTSS from baseline to 52 weeks between the etanercept 25 mg twice weekly group and Methotrexate group, assuming that the common standard deviation of the change of mTSS from baseline was 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — Based on rank transformed data: rank of change = rank baseline+treatment +pooled study center+prior methotrexate use. If overall treatment effect statistically significant, 3 pairwise comparisons conducted, otherwise no further testing was made
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model based on rank transformed data: rank of change = rank baseline + treatment + pooled study center + prior methotrexate use
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Test type: Non-Inferiority or Equivalence — An outcome showing that etanercept 10 mg was superior to methotrexate and the presence of numerical difference ≤0.5 mTSS units between etanercept 25 mg and etanercept 10 mg would support non-inferiority for the 2 etanercept treatments; p = 0.2634, ANCOVA — [p-value comment as in outcome 1, analysis 2]

2. Secondary Outcome: Change From Baseline in Modified Total Sharp Score (mTSS) at Week 24
Description: as for outcome 1
Time Frame: Week 24
Population: rITT
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 171 | 190 | 181
Scores on a scale | 5.11 (0.58) | 2.42 (0.48) | 1.74 (0.45)
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Test type: Superiority or Other; p = 0.2248, ANCOVA — [p-value comment as in outcome 1, analysis 2]

3. Secondary Outcome: Change From Baseline in Erosion Score at Weeks 24 and 52
Description: Joint erosion score: erosion severity in 44 joints (16 per hand, 6 per foot). Each joint scored according to surface area involved, from 0 (no erosion) to 5 (extensive bone loss from more than one half of articulating bone). Because each side of foot joint was graded, maximum erosion score for foot joint was 10. Thus, maximum erosion score was 280. Change = score at observation minus score at Baseline. An increase in score from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline, Week 24, and Week 52
Population: rITT
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 171 | 190 | 181
Scores on a scale
  Change at Week 24 | 2.90 (0.33) | 1.25 (0.29) | 1.12 (0.30)
  Change at Week 52 | 5.43 (0.64) | 2.75 (0.57) | 2.03 (0.48)
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.7260, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.5717, ANCOVA — [p-value comment as in outcome 1, analysis 2]

4. Secondary Outcome: Change From Baseline in Joint Space Narrowing (JSN) Score at Weeks 24 and 52
Description: JSN score: severity of JSN in 42 joints (15 per hand and 6 per foot), including subluxation, scored from 0 (no/normal JSN) to 4 (complete loss of joint space, bony ankylosis, or luxation). Maximum JSN score was 168. Change = scores at observation minus score at Baseline. An increase in score from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline, Week 24, and Week 52
Population: rITT
Measure: Mean (Standard Error); unit: Scores on a scale
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 171 | 190 | 181
Scores on a scale
  Change at Week 24 | 2.21 (0.34) | 1.18 (0.23) | 0.62 (0.20)
  Change at Week 52 | 4.39 (0.66) | 2.44 (0.42) | 1.31 (0.33)
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p = 0.0013, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.0186, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p = 0.0006, ANCOVA — [p-value comment as in outcome 1, analysis 2]
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.1123, ANCOVA — [p-value comment as in outcome 1, analysis 2]

5. Secondary Outcome: Percentage of Participants With no Progression of Joint Destruction at Week 52
Description: Absence of joint destruction defined by 3 categories (mTSS change <=0.5, <=3.0, and <smallest detectable difference [SDD] where SDDs were scores >3.0). mTSS = sum of erosion and JSN scores for 44 joints (16 per hand and 6 per foot). mTSS scores ranged from 0 (normal) to 448 (worst possible total score).
Time Frame: Baseline and Week 52
Population: rITT
Measure: Number; unit: Percentage of participants
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 171 | 190 | 181
Percentage of participants
  Progression ≤0.5 | 25.7 | 45.3 | 49.2
  Progression ≤3.0 | 46.8 | 64.2 | 68.0
  Progression ≤SDD | 81.9 | 88.9 | 94.5
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 52 for progression <=0.5; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — Stratified by pooled study center and prior methotrexate use
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 52 for progression <=0.5; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel — Stratified by pooled study center and prior methotrexate use
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52 for progression <=0.5; Test type: Superiority or Other; p = 0.3022, Cochran-Mantel-Haenszel — Stratified by pooled study center and prior methotrexate use
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 52 for progression <=3.0; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel — Stratified by pooled study center and prior methotrexate use
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 52 for progression <=3.0; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel — Stratified by pooled study center and prior methotrexate use
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52 for progression <=3.0; Test type: Superiority or Other; p = 0.3120, Cochran-Mantel-Haenszel — Stratified by pooled study center and prior methotrexate use
Statistical Analysis 7: Comparison: Methotrexate vs Etanercept 25 mg; Week 52 for progression <=SDD; Test type: Superiority or Other; p = 0.0010, Cochran-Mantel-Haenszel — Stratified by pooled study center and prior methotrexate use
Statistical Analysis 8: Comparison: Methotrexate vs Etanercept 10 mg; Week 52 for progression <=SDD; Test type: Superiority or Other; p = 0.0285, Cochran-Mantel-Haenszel — Stratified by pooled study center and prior methotrexate use
Statistical Analysis 9: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52 for progression <=SDD; Test type: Superiority or Other; p = 0.0433, Cochran-Mantel-Haenszel — Stratified by pooled study center and prior methotrexate use

6. Secondary Outcome: Change From Baseline in Swollen Joint Count at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Description: American College of Rheumatology (ACR) swollen joint count was an assessment of 68 joints. Joints classified as either swollen or not swollen. Change = scores at observation minus score at Baseline, and total possible scores ranged from -68 to 68. An increase in swollen joints from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: Modified ITT (mITT) population: participants who received at least 1 dose of the assigned test article; Last Observation Carried Forward (LOCF)
Measure: Mean (Standard Deviation); unit: Swollen Joints
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 176 | 192 | 182
Swollen Joints
  Baseline | 13.84 (7.81) | 14.23 (8.97) | 14.00 (8.80)
  Change at Week 2 | -3.39 (6.59) | -5.96 (6.94) | -5.02 (5.66)
  Change at Week 4 | -4.31 (6.68) | -7.03 (7.57) | -6.95 (6.35)
  Change at Week 8 | -5.76 (6.41) | -8.38 (7.77) | -7.91 (6.71)
  Change at Week 12 | -6.36 (6.97) | -9.05 (7.79) | -8.55 (6.72)
  Change at Week 16 | -6.59 (6.77) | -9.29 (7.93) | -8.78 (6.89)
  Change at Week 20 | -7.21 (7.47) | -9.68 (7.92) | -9.43 (7.45)
  Change at Week 24 | -7.06 (7.52) | -9.58 (7.98) | -9.57 (7.51)
  Change at Week 32 | -7.47 (7.74) | -9.89 (8.51) | -9.79 (7.62)
  Change at Week 40 | -7.93 (7.83) | -9.97 (8.53) | -10.05 (8.02)
  Change at Week 48 | -7.53 (8.26) | -9.87 (8.51) | -10.30 (8.41)
  Change at Week 52 | -7.53 (8.09) | -9.79 (8.58) | -10.49 (8.14)
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.0032, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.1224, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.8037, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 7: Comparison: Methotrexate vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 8: Comparison: Methotrexate vs Etanercept 10 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 9: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.5495, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 10: Comparison: Methotrexate vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 11: Comparison: Methotrexate vs Etanercept 10 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 12: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.4948, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 13: Comparison: Methotrexate vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 14: Comparison: Methotrexate vs Etanercept 10 mg; Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 15: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.4663, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 16: Comparison: Methotrexate vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 17: Comparison: Methotrexate vs Etanercept 10 mg; Week 20; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 18: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.9357, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 19: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 20: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 21: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.7439, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 22: Comparison: Methotrexate vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 23: Comparison: Methotrexate vs Etanercept 10 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 24: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p = 0.8611, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 25: Comparison: Methotrexate vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 26: Comparison: Methotrexate vs Etanercept 10 mg; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 27: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.6731, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 28: Comparison: Methotrexate vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 29: Comparison: Methotrexate vs Etanercept 10 mg; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 30: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.2616, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 31: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 32: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p = 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 33: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.1158, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment

7. Secondary Outcome: Change From Baseline in Number of Painful Joints on Pressure or on Motion at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Description: 71 joints assessed by the investigator using criteria based on pressure and joint manipulation. Change = scores at observation minus score at Baseline, and total possible scores ranged from -71 to 71. An increase in tender joint count from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Tender Joints
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 176 | 192 | 182
Tender Joints
  Baseline | 17.12 (10.78) | 16.30 (10.56) | 17.48 (11.21)
  Change at Week 2 | -3.41 (7.48) | -6.81 (7.67) | -7.73 (7.81)
  Change at Week 4 | -5.58 (8.34) | -7.74 (9.21) | -8.65 (7.75)
  Change at Week 8 | -6.83 (8.30) | -9.27 (9.50) | -10.86 (9.07)
  Change at Week 12 | -8.42 (9.08) | -9.94 (9.63) | -11.36 (9.20)
  Change at Week 16 | -8.82 (9.44) | -10.70 (9.79) | -11.81 (9.29)
  Change at Week 20 | -9.15 (9.93) | -10.86 (9.85) | -12.38 (10.10)
  Change at Week 24 | -9.47 (10.30) | -10.94 (9.64) | -12.48 (9.81)
  Change at Week 32 | -9.91 (10.56) | -10.93 (9.75) | -12.97 (10.14)
  Change at Week 40 | -9.97 (10.43) | -11.07 (10.32) | -12.73 (10.87)
  Change at Week 48 | -10.45 (10.69) | -10.78 (9.84) | -13.17 (11.20)
  Change at Week 52 | -10.27 (10.60) | -10.75 (9.99) | -13.23 (11.13)
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.4237, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 4; Test type: Superiority or Other; p = 0.0002, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.5738, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 7: Comparison: Methotrexate vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 8: Comparison: Methotrexate vs Etanercept 10 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 9: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.1606, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 10: Comparison: Methotrexate vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 11: Comparison: Methotrexate vs Etanercept 10 mg; Week 12; Test type: Superiority or Other; p = 0.0016, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 12: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.2412, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 13: Comparison: Methotrexate vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 14: Comparison: Methotrexate vs Etanercept 10 mg; Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 15: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.5882, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 16: Comparison: Methotrexate vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 17: Comparison: Methotrexate vs Etanercept 10 mg; Week 20; Test type: Superiority or Other; p = 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 18: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.2257, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 19: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 20: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p = 0.0003, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 21: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.2075, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 22: Comparison: Methotrexate vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 23: Comparison: Methotrexate vs Etanercept 10 mg; Week 32; Test type: Superiority or Other; p = 0.0050, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 24: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p = 0.0461, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 25: Comparison: Methotrexate vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.0002, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 26: Comparison: Methotrexate vs Etanercept 10 mg; Week 40; Test type: Superiority or Other; p = 0.0101, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 27: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.2351, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 28: Comparison: Methotrexate vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.0002, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 29: Comparison: Methotrexate vs Etanercept 10 mg; Week 48; Test type: Superiority or Other; p = 0.1179, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 30: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.0214, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 31: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 32: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p = 0.0790, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 33: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.0168, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment

8. Secondary Outcome: Change From Baseline in Physician's Global Assessment of Symptoms at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Description: Physician Global Assessment of symptoms, assessed using a 11-point rating scale, where 0=asymptomatic and 10=severe symptoms. Change = scores at observation minus score at Baseline. An increase in score from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 176 | 192 | 182
Scores on a scale
  Baseline | 6.34 (1.98) | 6.23 (1.79) | 6.20 (1.86)
  Week 2 | -1.23 (1.67) | -2.20 (1.71) | -2.25 (1.71)
  Week 4 | -1.66 (1.81) | -2.65 (1.91) | -2.67 (1.90)
  Week 8 | -2.13 (2.05) | -3.02 (1.89) | -3.14 (1.89)
  Week 12 | -2.43 (2.13) | -3.30 (2.04) | -3.34 (1.94)
  Week 16 | -2.51 (2.21) | -3.46 (2.02) | -3.53 (1.99)
  Week 20 | -2.54 (2.29) | -3.51 (2.07) | -3.76 (2.01)
  Week 24 | -2.60 (2.43) | -3.52 (2.22) | -3.76 (2.07)
  Week 32 | -2.70 (2.36) | -3.54 (2.24) | -3.94 (2.09)
  Week 40 | -2.63 (2.41) | -3.62 (2.28) | -3.97 (2.27)
  Week 48 | -2.70 (2.52) | -3.59 (2.45) | -4.03 (2.20)
  Week 52 | -2.72 (2.40) | -3.68 (2.42) | -4.07 (2.11)
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.6337, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.7407, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 7: Comparison: Methotrexate vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 8: Comparison: Methotrexate vs Etanercept 10 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 9: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.3473, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 10: Comparison: Methotrexate vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 11: Comparison: Methotrexate vs Etanercept 10 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 12: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.7529, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 13: Comparison: Methotrexate vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 14: Comparison: Methotrexate vs Etanercept 10 mg; Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 15: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.5216, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 16: Comparison: Methotrexate vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 17: Comparison: Methotrexate vs Etanercept 10 mg; Week 20; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 18: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.1078, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 19: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 20: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 21: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.1280, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 22: Comparison: Methotrexate vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 23: Comparison: Methotrexate vs Etanercept 10 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 24: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p = 0.0291, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 25: Comparison: Methotrexate vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 26: Comparison: Methotrexate vs Etanercept 10 mg; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 27: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.0729, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 28: Comparison: Methotrexate vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 29: Comparison: Methotrexate vs Etanercept 10 mg; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 30: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.0271, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 31: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 32: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 33: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.0453, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment

9. Secondary Outcome: Change From Baseline in Patient's Global Assessment at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Description: Patient's Global Assessment of symptoms, assessed using a 11-point rating scale, where 0=asymptomatic and 10=severe symptoms. Change = scores at observation minus score at Baseline. An increase in score from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 176 | 192 | 182
Scores on a scale
  Baseline | 6.01 (2.28) | 6.12 (2.17) | 5.95 (2.01)
  Change at Week 2 | -0.65 (1.95) | -1.81 (1.86) | -1.79 (1.82)
  Change at Week 4 | -1.11 (1.99) | -1.89 (2.06) | -1.91 (2.04)
  Change at Week 8 | -1.34 (2.31) | -2.37 (2.05) | -2.27 (2.13)
  Change at Week 12 | -1.63 (2.52) | -2.57 (2.22) | -2.38 (2.29)
  Change at Week 16 | -1.71 (2.45) | -2.55 (2.37) | -2.54 (2.40)
  Change at Week 20 | -1.85 (2.42) | -2.59 (2.36) | -2.69 (2.34)
  Change at Week 24 | -1.85 (2.66) | -2.65 (2.45) | -2.79 (2.45)
  Change at Week 32 | -1.89 (2.71) | -2.84 (2.44) | -2.92 (2.58)
  Change at Week 40 | -1.88 (2.68) | -2.89 (2.44) | -2.82 (2.67)
  Change at Week 48 | -1.97 (2.77) | -2.95 (2.46) | -2.98 (2.52)
  Change at Week 52 | -1.97 (2.70) | -3.04 (2.58) | -2.91 (2.60)
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.7488, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.5680, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 7: Comparison: Methotrexate vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 8: Comparison: Methotrexate vs Etanercept 10 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 9: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.9241, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 10: Comparison: Methotrexate vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 11: Comparison: Methotrexate vs Etanercept 10 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 12: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.7146, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 13: Comparison: Methotrexate vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 14: Comparison: Methotrexate vs Etanercept 10 mg; Week 16; Test type: Superiority or Other; p = 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 15: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.6574, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 16: Comparison: Methotrexate vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 17: Comparison: Methotrexate vs Etanercept 10 mg; Week 20; Test type: Superiority or Other; p = 0.0004, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 18: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.2936, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 19: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 20: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p = 0.0005, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 21: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.2179, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 22: Comparison: Methotrexate vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 23: Comparison: Methotrexate vs Etanercept 10 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 24: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p = 0.3704, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 25: Comparison: Methotrexate vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 26: Comparison: Methotrexate vs Etanercept 10 mg; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 27: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.8047, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 28: Comparison: Methotrexate vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 29: Comparison: Methotrexate vs Etanercept 10 mg; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 30: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.5277, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 31: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 32: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 33: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.9371, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment

10. Secondary Outcome: Change From Baseline in Mean Duration of Morning Stiffness at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Description: Morning stiffness in and around the joints lasting at least 1 hour before maximal improvement. Change = scores at observation minus score at Baseline. An increase in stiffness duration from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 176 | 192 | 182
Minutes
  Baseline | 204.74 (338.70) | 203.80 (304.92) | 223.48 (344.75)
  Change at Week 2 | -46.39 (250.13) | -98.73 (259.91) | -108.37 (256.49)
  Change at Week 4 | -34.43 (249.33) | -94.87 (280.56) | -107.09 (255.06)
  Change at Week 8 | -52.53 (247.74) | -122.13 (304.33) | -127.55 (279.88)
  Change at Week 12 | -73.48 (236.69) | -128.02 (309.89) | -129.74 (284.58)
  Change at Week 16 | -78.60 (252.64) | -136.18 (318.85) | -148.13 (304.03)
  Change at Week 20 | -87.11 (276.35) | -137.18 (320.34) | -153.01 (314.41)
  Change at Week 24 | -89.94 (295.48) | -137.72 (317.24) | -143.03 (332.16)
  Change at Week 32 | -95.32 (330.07) | -137.26 (332.50) | -163.64 (320.36)
  Change at Week 40 | -97.76 (332.93) | -142.06 (335.44) | -157.52 (336.53)
  Change at Week 48 | -99.38 (306.33) | -136.23 (333.45) | -163.03 (326.06)
  Change at Week 52 | -98.98 (303.71) | -124.86 (361.03) | -171.36 (322.43)
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.0027, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 2; Test type: Superiority or Other; p = 0.0015, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.8875, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.0015, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 4; Test type: Superiority or Other; p = 0.0011, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.9694, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 7: Comparison: Methotrexate vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.0020, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 8: Comparison: Methotrexate vs Etanercept 10 mg; Week 8; Test type: Superiority or Other; p = 0.0005, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 9: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.7271, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 10: Comparison: Methotrexate vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.0235, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 11: Comparison: Methotrexate vs Etanercept 10 mg; Week 12; Test type: Superiority or Other; p = 0.0061, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 12: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.6427, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 13: Comparison: Methotrexate vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.0036, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 14: Comparison: Methotrexate vs Etanercept 10 mg; Week 16; Test type: Superiority or Other; p = 0.0029, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 15: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.9713, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 16: Comparison: Methotrexate vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.0060, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 17: Comparison: Methotrexate vs Etanercept 10 mg; Week 20; Test type: Superiority or Other; p = 0.0060, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 18: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.9762, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 19: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.0554, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 20: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p = 0.0181, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 21: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.6642, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 22: Comparison: Methotrexate vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p = 0.0073, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 23: Comparison: Methotrexate vs Etanercept 10 mg; Week 32; Test type: Superiority or Other; p = 0.0290, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 24: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p = 0.5919, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 25: Comparison: Methotrexate vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.0371, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 26: Comparison: Methotrexate vs Etanercept 10 mg; Week 40; Test type: Superiority or Other; p = 0.0346, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 27: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.9955, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 28: Comparison: Methotrexate vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.0187, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 29: Comparison: Methotrexate vs Etanercept 10 mg; Week 48; Test type: Superiority or Other; p = 0.0645, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 30: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.5920, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 31: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.0095, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 32: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p = 0.2112, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 33: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.1649, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment

11. Secondary Outcome: Change From Baseline in Visual Analogue Scale for Pain (VAS-pain) at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Description: 100 millimeter (mm) line (VAS) marked by participant. Intensity of pain range (over past week): 0mm = no pain to 100mm = worst possible pain. Change = scores at observation minus score at Baseline. An increase in score from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 176 | 192 | 182
mm
  Baseline | 54.91 (23.62) | 54.37 (23.10) | 52.63 (21.54)
  Change at Week 2 | -5.98 (19.11) | -18.85 (19.76) | -18.67 (20.32)
  Change at Week 4 | -10.64 (21.45) | -18.18 (22.95) | -19.16 (21.86)
  Change at Week 8 | -13.48 (25.21) | -23.09 (22.37) | -22.46 (22.34)
  Change at Week 12 | -16.95 (25.09) | -24.70 (22.74) | -24.01 (22.70)
  Change at Week 16 | -17.97 (26.61) | -24.41 (24.53) | -25.63 (25.04)
  Change at Week 20 | -19.53 (24.67) | -25.39 (24.01) | -26.52 (24.58)
  Change at Week 24 | -19.53 (27.02) | -26.86 (24.37) | -26.73 (24.99)
  Change at Week 32 | -19.72 (27.01) | -28.68 (25.00) | -28.10 (25.85)
  Change at Week 40 | -19.68 (27.35) | -28.81 (26.09) | -27.17 (25.26)
  Change at Week 48 | -20.85 (28.08) | -28.28 (25.04) | -28.77 (25.50)
  Change at Week 52 | -20.03 (27.74) | -29.08 (25.85) | -28.34 (25.92)
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.8972, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.3736, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 7: Comparison: Methotrexate vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 8: Comparison: Methotrexate vs Etanercept 10 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 9: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.9324, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 10: Comparison: Methotrexate vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 11: Comparison: Methotrexate vs Etanercept 10 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 12: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.8982, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 13: Comparison: Methotrexate vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 14: Comparison: Methotrexate vs Etanercept 10 mg; Week 16; Test type: Superiority or Other; p = 0.0007, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 15: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.3180, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 16: Comparison: Methotrexate vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 17: Comparison: Methotrexate vs Etanercept 10 mg; Week 20; Test type: Superiority or Other; p = 0.0011, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 18: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.3302, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 19: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 20: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p = 0.0002, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 21: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.6563, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 22: Comparison: Methotrexate vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 23: Comparison: Methotrexate vs Etanercept 10 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 24: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p = 0.8894, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 25: Comparison: Methotrexate vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 26: Comparison: Methotrexate vs Etanercept 10 mg; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 27: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.7826, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 28: Comparison: Methotrexate vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 29: Comparison: Methotrexate vs Etanercept 10 mg; Week 48; Test type: Superiority or Other; p = 0.0003, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 30: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.5343, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 31: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 32: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 33: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.9313, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment

12. Secondary Outcome: Change From Baseline in VAS for Participant General Health at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Description: 100mm line (VAS) marked by participant. Participants asked, "In general how would you rate your health over the last 2-3 weeks?" 0mm=very well to 100mm=extremely bad. Change = scores at observation minus score at Baseline. An increase in score from baseline represented disease progression and/or joint worsening, no change represented halting of disease progression, and a decrease represented improvement.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 176 | 192 | 182
mm
  Baseline | 58.37 (24.04) | 58.71 (23.08) | 55.70 (21.68)
  Change at Week 2 | -8.06 (19.00) | -21.07 (20.39) | -20.27 (22.08)
  Change at Week 4 | -13.51 (21.35) | -20.65 (23.18) | -20.69 (22.47)
  Change at Week 8 | -15.59 (24.92) | -26.16 (23.39) | -25.57 (22.59)
  Change at Week 12 | -20.05 (25.50) | -28.08 (24.87) | -26.34 (23.27)
  Change at Week 16 | -20.89 (27.29) | -28.37 (26.15) | -27.30 (24.73)
  Change at Week 20 | -22.35 (25.37) | -29.51 (25.05) | -29.16 (24.79)
  Change at Week 24 | -21.78 (27.55) | -30.23 (25.23) | -29.52 (25.39)
  Change at Week 32 | -22.87 (27.60) | -31.92 (24.91) | -31.11 (25.86)
  Change at Week 40 | -22.69 (28.18) | -31.49 (27.26) | -30.36 (25.54)
  Change at Week 48 | -23.76 (29.21) | -32.15 (26.01) | -31.27 (25.42)
  Change at Week 52 | -23.34 (28.48) | -32.25 (27.02) | -31.08 (26.60)
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.8044, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 4; Test type: Superiority or Other; p = 0.0003, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.4652, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 7: Comparison: Methotrexate vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 8: Comparison: Methotrexate vs Etanercept 10 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 9: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.5612, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 10: Comparison: Methotrexate vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.0002, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 11: Comparison: Methotrexate vs Etanercept 10 mg; Week 12; Test type: Superiority or Other; p = 0.0002, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 12: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.9749, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 13: Comparison: Methotrexate vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 14: Comparison: Methotrexate vs Etanercept 10 mg; Week 16; Test type: Superiority or Other; p = 0.0004, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 15: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.7290, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 16: Comparison: Methotrexate vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 17: Comparison: Methotrexate vs Etanercept 10 mg; Week 20; Test type: Superiority or Other; p = 0.0003, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 18: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.5004, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 19: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 20: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 21: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.5727, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 22: Comparison: Methotrexate vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 23: Comparison: Methotrexate vs Etanercept 10 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 24: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p = 0.6713, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 25: Comparison: Methotrexate vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 26: Comparison: Methotrexate vs Etanercept 10 mg; Week 40; Test type: Superiority or Other; p = 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 27: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.7663, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 28: Comparison: Methotrexate vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 29: Comparison: Methotrexate vs Etanercept 10 mg; Week 48; Test type: Superiority or Other; p = 0.0002, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 30: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.7073, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 31: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 32: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p = 0.0001, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 33: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.7973, ANCOVA — P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment

13. Secondary Outcome: Change From Baseline in Health Assessment Questionnaire-Disability Index (HAQ-DI) Score at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Description: HAQ-DI: participant-reported assessment of ability to perform tasks: 1) dress/groom; 2) arise; 3) eat; 4) walk; 5) reach; 6) grip; 7) hygiene; and 8) common activities over past week. Each item scored on 4-point Likert scale from 0 to 3: 0=no difficulty; 1=some difficulty; 2=much difficulty; 3=unable to do. Change = scores at observation minus score at Baseline and total possible scores ranged from -3 to 3. An increase in score from baseline represented disease progression and/or joint worsening and a decrease represented improvement.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 176 | 192 | 182
Scores on a scale
  Baseline | 1.01 (0.65) | 1.17 (0.66) | 1.06 (0.67)
  Change at Week 2 | -0.06 (0.36) | -0.30 (0.34) | -0.34 (0.41)
  Change at Week 4 | -0.12 (0.44) | -0.33 (0.39) | -0.40 (0.43)
  Change at Week 8 | -0.21 (0.49) | -0.46 (0.45) | -0.48 (0.46)
  Change at Week 12 | -0.29 (0.54) | -0.51 (0.48) | -0.52 (0.49)
  Change at Week 16 | -0.30 (0.55) | -0.52 (0.51) | -0.54 (0.52)
  Change at Week 20 | -0.32 (0.58) | -0.49 (0.53) | -0.57 (0.54)
  Change at Week 24 | -0.33 (0.62) | -0.54 (0.52) | -0.59 (0.55)
  Change at Week 32 | -0.33 (0.64) | -0.56 (0.52) | -0.59 (0.59)
  Change at Week 40 | -0.35 (0.64) | -0.56 (0.55) | -0.60 (0.60)
  Change at Week 48 | -0.34 (0.65) | -0.57 (0.57) | -0.59 (0.57)
  Change at Week 52 | -0.35 (0.64) | -0.56 (0.56) | -0.58 (0.59)
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.1053, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.0144, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 7: Comparison: Methotrexate vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 8: Comparison: Methotrexate vs Etanercept 10 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 9: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.1851, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 10: Comparison: Methotrexate vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 11: Comparison: Methotrexate vs Etanercept 10 mg; Week 12; Test type: Superiority or Other; p = 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 12: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.2883, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 13: Comparison: Methotrexate vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 14: Comparison: Methotrexate vs Etanercept 10 mg; Week 16; Test type: Superiority or Other; p = 0.0007, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 15: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.2221, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 16: Comparison: Methotrexate vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 17: Comparison: Methotrexate vs Etanercept 10 mg; Week 20; Test type: Superiority or Other; p = 0.0147, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 18: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.0201, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 19: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 20: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p = 0.0036, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 21: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.0789, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 22: Comparison: Methotrexate vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 23: Comparison: Methotrexate vs Etanercept 10 mg; Week 32; Test type: Superiority or Other; p = 0.0008, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 24: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p = 0.1903, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 25: Comparison: Methotrexate vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 26: Comparison: Methotrexate vs Etanercept 10 mg; Week 40; Test type: Superiority or Other; p = 0.0048, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 27: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.1059, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 28: Comparison: Methotrexate vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 29: Comparison: Methotrexate vs Etanercept 10 mg; Week 48; Test type: Superiority or Other; p = 0.0018, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 30: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.2589, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 31: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 32: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p = 0.0040, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 33: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.2326, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment

14. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 20% (ACR20) Response
Description: ACR20 response: greater than or equal to (≥) 20 percent (%) improvement in tender joint count; ≥ 20% improvement in swollen joint count; and ≥ 20% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the Health Assessment Questionnaire [HAQ]); and C-Reactive Protein (CRP).
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: mITT; LOCF
Measure: Number; unit: Percentage of participants
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 176 | 192 | 182
Percentage of participants
  Week 2 | 16.1 | 54.0 | 49.4
  Week 4 | 27.3 | 55.5 | 56.9
  Week 8 | 43.2 | 68.1 | 68.7
  Week 12 | 48.3 | 70.2 | 77.5
  Week 16 | 51.7 | 73.8 | 75.3
  Week 20 | 58.5 | 75.4 | 78.6
  Week 24 | 56.3 | 77.0 | 77.5
  Week 32 | 58.0 | 79.1 | 80.8
  Week 40 | 59.7 | 78.5 | 75.3
  Week 48 | 59.1 | 76.4 | 79.7
  Week 52 | 62.5 | 75.9 | 78.6
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 2; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.4751, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 4; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.4653, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 7: Comparison: Methotrexate vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 8: Comparison: Methotrexate vs Etanercept 10 mg; Week 8; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 9: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.7953, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 10: Comparison: Methotrexate vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 11: Comparison: Methotrexate vs Etanercept 10 mg; Week 12; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 12: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.0848, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 13: Comparison: Methotrexate vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 14: Comparison: Methotrexate vs Etanercept 10 mg; Week 16; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 15: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.6112, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 16: Comparison: Methotrexate vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 17: Comparison: Methotrexate vs Etanercept 10 mg; Week 20; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 18: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.3671, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 19: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 20: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 21: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.7618, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 22: Comparison: Methotrexate vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 23: Comparison: Methotrexate vs Etanercept 10 mg; Week 32; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 24: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p = 0.4358, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 25: Comparison: Methotrexate vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.0008, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 26: Comparison: Methotrexate vs Etanercept 10 mg; Week 40; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 27: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.6267, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 28: Comparison: Methotrexate vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 29: Comparison: Methotrexate vs Etanercept 10 mg; Week 48; Test type: Superiority or Other; p = 0.0004, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 30: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.3564, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 31: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.0007, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 32: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p = 0.0035, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 33: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.4749, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use

15. Secondary Outcome: Percentage of Participants With an ACR50 Response
Description: ACR50 response: ≥ 50% improvement in tender joint count; ≥ 50% improvement in swollen joint count; and ≥ 50% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: mITT; LOCF
Measure: Number; unit: Percentage of participants
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 176 | 192 | 182
Percentage of participants
  Week 2 | 2.3 | 14.7 | 16.0
  Week 4 | 4.0 | 28.1 | 22.5
  Week 8 | 15.3 | 38.5 | 35.7
  Week 12 | 23.9 | 47.4 | 42.3
  Week 16 | 26.1 | 50.0 | 44.0
  Week 20 | 30.7 | 50.0 | 50.5
  Week 24 | 32.4 | 53.6 | 54.4
  Week 32 | 34.7 | 60.4 | 59.3
  Week 40 | 36.9 | 60.4 | 58.8
  Week 48 | 39.2 | 57.3 | 57.7
  Week 52 | 36.9 | 59.4 | 62.1
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 2; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.4376, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 4; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.3947, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 7: Comparison: Methotrexate vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 8: Comparison: Methotrexate vs Etanercept 10 mg; Week 8; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 9: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.7378, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 10: Comparison: Methotrexate vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 11: Comparison: Methotrexate vs Etanercept 10 mg; Week 12; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 12: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.5680, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 13: Comparison: Methotrexate vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 14: Comparison: Methotrexate vs Etanercept 10 mg; Week 16; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 15: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.3978, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 16: Comparison: Methotrexate vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 17: Comparison: Methotrexate vs Etanercept 10 mg; Week 20; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 18: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.7229, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 19: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 20: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 21: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.7236, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 22: Comparison: Methotrexate vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 23: Comparison: Methotrexate vs Etanercept 10 mg; Week 32; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 24: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p = 0.9719, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 25: Comparison: Methotrexate vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 26: Comparison: Methotrexate vs Etanercept 10 mg; Week 40; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 27: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.9349, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 28: Comparison: Methotrexate vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 29: Comparison: Methotrexate vs Etanercept 10 mg; Week 48; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 30: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.7226, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 31: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 32: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 33: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.5512, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use

16. Secondary Outcome: Percentage of Participants With an ACR70 Response
Description: ACR70 response: ≥ 70% improvement in tender joint count; ≥ 70% improvement in swollen joint count; and ≥ 70% improvement in at least 3 of 5 remaining ACR core measures: participant assessment of pain; participant global assessment of disease activity; physician global assessment of disease activity; self-assessed disability (disability index of the HAQ); and CRP.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: mITT; LOCF
Measure: Number; unit: Percentage of participants
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 176 | 192 | 182
Percentage of participants
  Week 2 | 0 | 4.2 | 3.8
  Week 4 | 0.6 | 7.8 | 8.2
  Week 8 | 2.8 | 15.1 | 11.0
  Week 12 | 9.7 | 21.9 | 15.4
  Week 16 | 9.7 | 17.7 | 18.7
  Week 20 | 13.1 | 25.0 | 25.3
  Week 24 | 11.9 | 25.5 | 25.8
  Week 32 | 11.9 | 28.1 | 31.3
  Week 40 | 14.8 | 31.3 | 35.7
  Week 48 | 18.2 | 34.4 | 36.3
  Week 52 | 15.9 | 33.9 | 36.3
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.0162, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 2; Test type: Superiority or Other; p = 0.0035, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.8928, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 4; Test type: Superiority or Other; p = 0.0007, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.6348, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 7: Comparison: Methotrexate vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.0026, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 8: Comparison: Methotrexate vs Etanercept 10 mg; Week 8; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 9: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.4629, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 10: Comparison: Methotrexate vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.0841, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 11: Comparison: Methotrexate vs Etanercept 10 mg; Week 12; Test type: Superiority or Other; p = 0.0007, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 12: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.1957, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 13: Comparison: Methotrexate vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.0093, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 14: Comparison: Methotrexate vs Etanercept 10 mg; Week 16; Test type: Superiority or Other; p = 0.0326, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 15: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.7426, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 16: Comparison: Methotrexate vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.0013, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 17: Comparison: Methotrexate vs Etanercept 10 mg; Week 20; Test type: Superiority or Other; p = 0.0015, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 18: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.6552, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 19: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.0005, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 20: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p = 0.0004, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 21: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.6294, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 22: Comparison: Methotrexate vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 23: Comparison: Methotrexate vs Etanercept 10 mg; Week 32; Test type: Superiority or Other; p = 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 24: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p = 0.4652, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 25: Comparison: Methotrexate vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 26: Comparison: Methotrexate vs Etanercept 10 mg; Week 40; Test type: Superiority or Other; p = 0.0002, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 27: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.2233, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 28: Comparison: Methotrexate vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 29: Comparison: Methotrexate vs Etanercept 10 mg; Week 48; Test type: Superiority or Other; p = 0.0003, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 30: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.6772, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 31: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 32: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use
Statistical Analysis 33: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.6160, Cochran-Mantel-Haenszel; Stratified by pooled study center and prior methotrexate use

17. Secondary Outcome: Change From Baseline in Disease Activity Score (DAS) at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Description: DAS: weighted calculation of joint tenderness score (Ritchie Articular Index[RAI]), swollen joint count of 44 joints, natural logarithm (ln) of erythrocyte sedimentation rate (ESR) in millimeters per hour (mm/hr), and general health (GH) using VAS. RAI defined as sum of 26 possible 0 to 3 tender scores. DAS = 0.53938 square root (√) (RAI) + 0.06465 (swollen joint count) + 0.330 (ln ESR) + 0.00722 (GH). Change from baseline = DAS at Week x minus Baseline DAS. Total DAS scores could range from 10 (worse outcome) to 0 (better outcome).
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 176 | 192 | 182
Scores on a scale
  Baseline | 4.07 (0.95) | 4.03 (0.89) | 4.05 (0.88)
  Change at Week 2 | -0.48 (0.64) | -1.09 (0.72) | -1.05 (0.70)
  Change at Week 4 | -0.69 (0.67) | -1.26 (0.90) | -1.26 (0.80)
  Change at Week 8 | -0.93 (0.79) | -1.48 (0.88) | -1.54 (0.86)
  Change at Week 12 | -1.12 (0.93) | -1.66 (0.97) | -1.65 (0.83)
  Change at Week 16 | -1.19 (0.98) | -1.69 (0.98) | -1.72 (0.88)
  Change at Week 20 | -1.28 (1.00) | -1.74 (0.97) | -1.80 (0.93)
  Change at Week 24 | -1.31 (1.09) | -1.77 (1.03) | -1.87 (0.98)
  Change at Week 32 | -1.37 (1.08) | -1.80 (1.02) | -1.95 (1.01)
  Change at Week 40 | -1.36 (1.08) | -1.90 (1.10) | -1.97 (1.02)
  Change at Week 48 | -1.46 (1.17) | -1.86 (1.13) | -2.02 (1.04)
  Change at Week 52 | -1.42 (1.14) | -1.86 (1.14) | -2.01 (1.06)
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.4929, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.9693, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 7: Comparison: Methotrexate vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 8: Comparison: Methotrexate vs Etanercept 10 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 9: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.4139, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 10: Comparison: Methotrexate vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 11: Comparison: Methotrexate vs Etanercept 10 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 12: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.8905, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 13: Comparison: Methotrexate vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 14: Comparison: Methotrexate vs Etanercept 10 mg; Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 15: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.6877, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 16: Comparison: Methotrexate vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 17: Comparison: Methotrexate vs Etanercept 10 mg; Week 20; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 18: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.4511, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 19: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 20: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 21: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.2786, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 22: Comparison: Methotrexate vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 23: Comparison: Methotrexate vs Etanercept 10 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 24: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p = 0.1230, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 25: Comparison: Methotrexate vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 26: Comparison: Methotrexate vs Etanercept 10 mg; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 27: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.5061, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 28: Comparison: Methotrexate vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 29: Comparison: Methotrexate vs Etanercept 10 mg; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 30: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.1354, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 31: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 32: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 33: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.1734, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment

18. Secondary Outcome: Change From Baseline in Disease Activity Score in 28 Joints (DAS28) at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Description: DAS based on 28 painful joint counts, 28 swollen joint counts, ESR, and GH. DAS28 score calculated as 0.56 √ (28 painful joint count) + 0.28 √ (28 swollen joint count) + 0.70 (ln ESR mm/hr) + 0.014 GH. Change from baseline = DAS at Week x minus Baseline DAS. Total DAS scores could range from 10 (worse outcome) to 0 (better outcome).
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 176 | 192 | 182
Scores on a scale
  Baseline | 5.84 (1.13) | 5.75 (1.17) | 5.82 (1.02)
  Change at Week 2 | -0.52 (0.75) | -1.32 (0.86) | -1.38 (0.88)
  Change at Week 4 | -0.77 (0.83) | -1.51 (1.05) | -1.60 (1.02)
  Change at Week 8 | -1.08 (0.99) | -1.79 (1.05) | -1.96 (1.11)
  Change at Week 12 | -1.33 (1.16) | -2.00 (1.15) | -2.09 (1.13)
  Change at Week 16 | -1.42 (1.24) | -2.08 (1.22) | -2.20 (1.17)
  Change at Week 20 | -1.54 (1.28) | -2.13 (1.24) | -2.31 (1.21)
  Change at Week 24 | -1.54 (1.34) | -2.20 (1.31) | -2.36 (1.27)
  Change at Week 32 | -1.63 (1.34) | -2.22 (1.29) | -2.45 (1.31)
  Change at Week 40 | -1.61 (1.36) | -2.31 (1.44) | -2.45 (1.33)
  Change at Week 48 | -1.75 (1.48) | -2.28 (1.51) | -2.51 (1.37)
  Change at Week 52 | -1.71 (1.44) | -2.25 (1.55) | -2.50 (1.38)
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.6417, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.4698, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 7: Comparison: Methotrexate vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 8: Comparison: Methotrexate vs Etanercept 10 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 9: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.1214, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 10: Comparison: Methotrexate vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 11: Comparison: Methotrexate vs Etanercept 10 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 12: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.4654, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 13: Comparison: Methotrexate vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 14: Comparison: Methotrexate vs Etanercept 10 mg; Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 15: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.4006, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 16: Comparison: Methotrexate vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 17: Comparison: Methotrexate vs Etanercept 10 mg; Week 20; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 18: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.1636, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 19: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 20: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 21: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.2635, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 22: Comparison: Methotrexate vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 23: Comparison: Methotrexate vs Etanercept 10 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 24: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p = 0.0965, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 25: Comparison: Methotrexate vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 26: Comparison: Methotrexate vs Etanercept 10 mg; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 27: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.4437, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 28: Comparison: Methotrexate vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 29: Comparison: Methotrexate vs Etanercept 10 mg; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 30: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.1663, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 31: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 32: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 33: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.1049, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment

19. Secondary Outcome: Change From Baseline in C-reactive Protein (CRP) at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Description: CRP: marker of inflammation. Higher level consistent with inflammation. Normal CRP range: 0 to 1.0 milligrams per deciliter (mg/dL).
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 176 | 192 | 182
mg/dL
  Baseline | 21.13 (22.30) | 22.86 (29.77) | 22.09 (24.17)
  Change at Week 2 | -3.08 (13.08) | -13.41 (19.53) | -15.62 (17.70)
  Change at Week 4 | -3.25 (15.82) | -11.05 (17.73) | -13.33 (16.58)
  Change at Week 8 | -4.19 (17.81) | -13.18 (20.74) | -15.17 (19.05)
  Change at Week 12 | -7.30 (18.00) | -13.04 (20.48) | -14.87 (20.36)
  Change at Week 16 | -6.51 (19.28) | -13.31 (20.73) | -15.15 (20.82)
  Change at Week 20 | -7.18 (21.29) | -12.21 (22.31) | -15.86 (20.23)
  Change at Week 24 | -6.31 (21.74) | -13.69 (21.26) | -16.28 (21.25)
  Change at Week 32 | -6.41 (21.68) | -13.45 (21.76) | -16.10 (21.38)
  Change at Week 40 | -6.23 (22.16) | -13.13 (22.47) | -15.38 (21.80)
  Change at Week 48 | -6.34 (22.18) | -13.01 (22.03) | -15.73 (22.44)
  Change at Week 52 | -5.20 (22.55) | -12.90 (22.96) | -15.08 (22.29)
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.0442, ANCOVA; P-values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.0681, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 7: Comparison: Methotrexate vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 8: Comparison: Methotrexate vs Etanercept 10 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 9: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.0966, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 10: Comparison: Methotrexate vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 11: Comparison: Methotrexate vs Etanercept 10 mg; Week 12; Test type: Superiority or Other; p = 0.0006, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 12: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.1242, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 13: Comparison: Methotrexate vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 14: Comparison: Methotrexate vs Etanercept 10 mg; Week 16; Test type: Superiority or Other; p < 0.001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 15: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.1521, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 16: Comparison: Methotrexate vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 17: Comparison: Methotrexate vs Etanercept 10 mg; Week 20; Test type: Superiority or Other; p = 0.0070, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 18: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.0140, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 19: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 20: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 21: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.0815, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 22: Comparison: Methotrexate vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 23: Comparison: Methotrexate vs Etanercept 10 mg; Week 32; Test type: Superiority or Other; p = 0.0002, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 24: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p = 0.0886, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 25: Comparison: Methotrexate vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 26: Comparison: Methotrexate vs Etanercept 10 mg; Week 40; Test type: Superiority or Other; p = 0.0003, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 27: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.1488, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 28: Comparison: Methotrexate vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 29: Comparison: Methotrexate vs Etanercept 10 mg; Week 48; Test type: Superiority or Other; p = 0.0006, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 30: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.0979, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 31: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 32: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p = 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment
Statistical Analysis 33: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.1740, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior methotrexate use + treatment

20. Secondary Outcome: Change From Baseline in Erythrocyte Sedimentation Rate (ESR) at Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Description: ESR: laboratory test that provided a non-specific measure of inflammation. The test assessed the rate at which red blood cells fell in a test tube and was measured in mm/hour. Normal range: 0-30mm/h. Higher rate consistent with inflammation.
Time Frame: Baseline and Weeks 2, 4, 8, 12, 16, 20, 24, 32, 40, 48, and 52
Population: mITT; LOCF
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 176 | 192 | 182
mm/hr
  Baseline | 42.55 (28.24) | 42.00 (29.44) | 43.66 (27.64)
  Change at Week 2 | -1.86 (10.65) | -13.67 (13.07) | -16.91 (15.01)
  Change at Week 4 | -2.92 (11.78) | -13.26 (14.94) | -16.62 (16.03)
  Change at Week 8 | -5.50 (16.89) | -13.99 (17.39) | -18.01 (17.83)
  Change at Week 12 | -8.89 (17.38) | -15.18 (17.63) | -18.98 (19.04)
  Change at Week 16 | -8.56 (18.73) | -15.45 (18.54) | -19.78 (20.32)
  Change at Week 20 | -10.56 (20.45) | -15.68 (19.15) | -19.40 (20.18)
  Change at Week 24 | -9.88 (20.15) | -16.52 (20.09) | -20.01 (20.86)
  Change at Week 32 | -9.92 (20.51) | -16.06 (21.14) | -20.16 (21.54)
  Change at Week 40 | -9.33 (20.50) | -15.93 (21.47) | -18.28 (21.81)
  Change at Week 48 | -10.70 (20.93) | -15.61 (23.07) | -19.25 (21.77)
  Change at Week 52 | -10.22 (21.69) | -14.79 (23.06) | -18.85 (21.67)
Statistical Analysis 1: Comparison: Methotrexate vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior Methotrexate use + treatment
Statistical Analysis 2: Comparison: Methotrexate vs Etanercept 10 mg; Week 2; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 3: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 2; Test type: Superiority or Other; p = 0.0274, ANCOVA — p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 4: Comparison: Methotrexate vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 5: Comparison: Methotrexate vs Etanercept 10 mg; Week 4; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 6: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 4; Test type: Superiority or Other; p = 0.0344, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 7: Comparison: Methotrexate vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 8: Comparison: Methotrexate vs Etanercept 10 mg; Week 8; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 9: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 8; Test type: Superiority or Other; p = 0.0293, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 10: Comparison: Methotrexate vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 11: Comparison: Methotrexate vs Etanercept 10 mg; Week 12; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 12: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 12; Test type: Superiority or Other; p = 0.0452, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 13: Comparison: Methotrexate vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 14: Comparison: Methotrexate vs Etanercept 10 mg; Week 16; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 15: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 16; Test type: Superiority or Other; p = 0.0313, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 16: Comparison: Methotrexate vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 17: Comparison: Methotrexate vs Etanercept 10 mg; Week 20; Test type: Superiority or Other; p = 0.0019, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 18: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 20; Test type: Superiority or Other; p = 0.0781, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 19: Comparison: Methotrexate vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 20: Comparison: Methotrexate vs Etanercept 10 mg; Week 24; Test type: Superiority or Other; p = 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 21: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 24; Test type: Superiority or Other; p = 0.1279, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 22: Comparison: Methotrexate vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 23: Comparison: Methotrexate vs Etanercept 10 mg; Week 32; Test type: Superiority or Other; p = 0.0004, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 24: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 32; Test type: Superiority or Other; p = 0.0807, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 25: Comparison: Methotrexate vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 26: Comparison: Methotrexate vs Etanercept 10 mg; Week 40; Test type: Superiority or Other; p = 0.0002, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 27: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 40; Test type: Superiority or Other; p = 0.4180, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 28: Comparison: Methotrexate vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 29: Comparison: Methotrexate vs Etanercept 10 mg; Week 48; Test type: Superiority or Other; p = 0.0061, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 30: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 48; Test type: Superiority or Other; p = 0.1615, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 31: Comparison: Methotrexate vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p < 0.0001, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 32: Comparison: Methotrexate vs Etanercept 10 mg; Week 52; Test type: Superiority or Other; p = 0.0130, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment
Statistical Analysis 33: Comparison: Etanercept 10 mg vs Etanercept 25 mg; Week 52; Test type: Superiority or Other; p = 0.0948, ANCOVA; p-Values from ANCOVA model: change = baseline + pooled study center + prior MTX use + treatment

21. Other Pre Specified Outcome: Comparison of Etanercept Serum Concentrations Between the 10 mg and 25 mg Etanercept Doses
Time Frame: Weeks 12, 24, 52
Population: mITT; n = evaluable participants at the specified time point.
Measure: Mean (Standard Error); unit: nanograms per milliliter (ng/mL)
Arm/Group | Etanercept 10 mg | Etanercept 25 mg
Number analyzed (Participants) | 179 | 171
nanograms per milliliter (ng/mL)
  Week 12 (n=179, 164) | 1012 (30.3) | 2490 (79.6)
  Week 24 (n=171, 171) | 1094 (32.2) | 2500 (79.3)
  Week 52 (n=158, 149) | 1097 (34.4) | 2754 (136)

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious AE (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Methotrexate | Etanercept 10 mg | Etanercept 25 mg
Serious Adverse Events (participants affected / at risk) | 10/176 | 8/192 | 11/182
Other Adverse Events (participants affected / at risk) | 92/176 | 106/192 | 102/182
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=176) | Etanercept 10 mg (N=192) | Etanercept 25 mg (N=182)
Sudden hearing loss (Ear and labyrinth disorders) | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 0 | 1
Thyroiditis subacute (Endocrine disorders) | 0 | 0 | 1
Retinal detachment (Eye disorders) | 0 | 1 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Ulna fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Occipital neuralgia (Nervous system disorders) | 0 | 0 | 1
Abortion (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=176) | Etanercept 10 mg (N=192) | Etanercept 25 mg (N=182)
Palpitations (Cardiac disorders) | 4 | 0 | 2
Vertigo (Ear and labyrinth disorders) | 0 | 5 | 1
Conjunctivitis allergic (Eye disorders) | 2 | 0 | 4
Abdominal discomfort (Gastrointestinal disorders) | 4 | 6 | 0
Abdominal pain upper (Gastrointestinal disorders) | 5 | 3 | 3
Constipation (Gastrointestinal disorders) | 9 | 6 | 7
Diarrhoea (Gastrointestinal disorders) | 5 | 5 | 10
Gastritis (Gastrointestinal disorders) | 6 | 3 | 1
Nausea (Gastrointestinal disorders) | 7 | 4 | 1
Stomatitis (Gastrointestinal disorders) | 8 | 8 | 3
Vomiting (Gastrointestinal disorders) | 1 | 3 | 4
Pyrexia (General disorders) | 6 | 2 | 8
Hepatic function abnormal (Hepatobiliary disorders) | 6 | 5 | 3
Contusion (Injury, poisoning and procedural complications) | 4 | 4 | 8
Alanine aminotransferase increased (Investigations) | 22 | 12 | 10
Aspartate aminotransferase increased (Investigations) | 18 | 8 | 8
Blood alkaline phosphatase increased (Investigations) | 3 | 2 | 5
Blood pressure increased (Investigations) | 3 | 3 | 4
Blood urine present (Investigations) | 2 | 5 | 2
Transaminases increased (Investigations) | 8 | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 2 | 1
Dizziness (Nervous system disorders) | 1 | 6 | 3
Headache (Nervous system disorders) | 4 | 5 | 9
Insomnia (Psychiatric disorders) | 9 | 9 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 6
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 3 | 6 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 2 | 4
Dermatitis contact (Skin and subcutaneous tissue disorders) | 4 | 3 | 4
Eczema (Skin and subcutaneous tissue disorders) | 8 | 7 | 8
Erythema (Skin and subcutaneous tissue disorders) | 1 | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 12 | 5
Rash (Skin and subcutaneous tissue disorders) | 8 | 10 | 10
Urticaria (Skin and subcutaneous tissue disorders) | 2 | 4 | 1
Hypertension (Vascular disorders) | 2 | 4 | 4
Dental caries (Gastrointestinal disorders) | 3 | 4 | 8
Periodontitis (Gastrointestinal disorders) | 0 | 1 | 5
Bronchitis (Infections and infestations) | 5 | 5 | 6
Cystitis (Infections and infestations) | 6 | 4 | 9
Gastroenteritis (Infections and infestations) | 5 | 1 | 1
Hordeolum (Infections and infestations) | 1 | 2 | 4
Influenza (Infections and infestations) | 6 | 4 | 1
Nasopharyngitis (Infections and infestations) | 43 | 45 | 37
Oral herpes (Infections and infestations) | 2 | 6 | 2
Otitis media (Infections and infestations) | 1 | 4 | 0
Pharyngitis (Infections and infestations) | 12 | 18 | 15
Pneumonia (Infections and infestations) | 0 | 5 | 2
Upper respiratory tract infection (Infections and infestations) | 20 | 20 | 21

LIMITATIONS AND CAVEATS:
Total Sharp Score and modified total Sharp Score were used interchangeably in the protocol and meant the same thing. In the statistical analysis plan and study results, mTSS was used consistently.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Wyeth has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.